CLINICAL TRIAL: NCT06003959
Title: The Effect of Breastfeeding Support System on Breast Milk Quantity and Mother-Infant Bonding in Preterm Infants: a Randomized Controlled Study
Brief Title: The Effect of Breastfeeding Support System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sümeyye EKİCİ, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sumeyye
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-08

CONDITIONS: Preterm; Breastfeeding; Breast Milk; Breastfeeding Support System
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breastfeeding Support System (Experimental): The intervention group was given breastfeeding support system care
  Interventions: Other: Routine nursing care; Other: breastfeeding support system
- Control group (No Intervention): Routine nursing care was given to the pretrms in this groups without any breastfeeding support system care

INTERVENTIONS:
Other: Routine nursing care — Preterm infants in the control group did not receive any intervention other than the routine feeding protocol applied in the clinic.
  Arms: Breastfeeding Support System
Other: breastfeeding support system — The body weight of preterm infants in the experimental group was measured and recorded each morning before their first feeding. Mothers of these infants were asked to complete the Mother-Infant Attachment Scale (MIAS) prior to the procedure. The physician determined the appropriate amount of breast milk the infant should receive during feeding. Before each feeding, the neonatal nurse ensured the sterile preparation of the milk and transferred it to the Breastfeeding Support System. The mothers were then prepared for the procedure, with the neonatal nurse explaining how the breastfeeding support system worked. Once both the mother and baby were ready, the baby was placed at the mother's breast. After feeding, the mothers were asked to complete the MIAS again.
  Arms: Breastfeeding Support System

SUMMARY:
This study aimed to examine the impact of a breastfeeding support system on breast milk production and mother-infant bonding in preterm infants. The sample included 70 preterm infants and their mothers, divided into two groups: 35 in the control group and 35 in the experimental group, all of whom met the study criteria.

ELIGIBILITY:
Inclusion Criteria:

For the infant:

Gestational age between 30 and 34 weeks Birth weight of 1000 g or more

For the mother:

Age over 18, literate, and able to speak Turkish Willingness to breastfeed and no chronic illness preventing breastfeeding

Exclusion Criteria:

Infants without identification Infants with unstable vital signs Mothers with conditions that prevent breastfeeding

Ages: 30 Months to 34 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mother-Infant Attachment Scale | up to 6 months
  The Turkish validity and reliability of this scale, originally developed by Taylor et al. in 2005, were established by Aydemir Karakulak and Alparslan in 2016. It can be easily and quickly administered by the mother from the first day after birth. The scale consists of 8 items with a four-point Likert-type format. Scores range from 0 to 24, with higher scores indicating a potential attachment issue between the mother and infant.

CONTACTS AND LOCATIONS:
Locations (1):
- Sümeyye EKİCİ, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No